CLINICAL TRIAL: NCT04482127
Title: Post-extraction Volumetric Analysis of Alveolar Ridge Contour Using Subepithelial Connective Tissue Graft in Esthetic Zone: A Randomized Controlled Clinical Trial
Brief Title: Volumetric Analysis of Alveolar Ridge Contour Using Sub-epithelial Connective Tissue Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gamal A Aziz, Masters Student at Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PER 632
Record Dates: First submitted 2020-04-27; First posted 2020-07-22 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Alveolar Ridge Collapse

STUDY DESIGN:
Intervention Model Description: Group A will receive atraumatic extraction and soft tissue augmentation using SCTG harvested from palatal tissue by single line incision technique (Hürzeler and Weng, 1999) blade will be oriented perpendicular to the palatal tissue surface. A single incision will be made down to the bone in a horizontal direction approximately 2 to 3 mm apical to the gingival margin of the maxillary teeth. A partial thickness dissection will then be made within the single incision, leaving an adequate thickness of the palatal flap intact to minimize the chance of sloughing of the overlying tissue. Careful manipulation of the graft with tissue forceps will be required and care must be taken to prevent compression or tearing of the graft.
  Group B will receive atraumatic extraction with no soft tissue augmentation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SubEpithelial connective graft (Experimental): SCTG harvested from palatal tissue by single line incision technique, blade will be oriented perpendicular to the palatal tissue surface. A single incision will be made down to the bone in a horizontal direction approximately 2 to 3 mm apical to the gingival margin of the maxillary teeth. A partial thickness dissection will then be made within the single incision, leaving an adequate thickness of the palatal flap intact to minimize the chance of sloughing of the overlying tissue. Careful manipulation of the graft with tissue forceps will be required and care must be taken to prevent compression or tearing of the graft.
  The fatty tissue (yellow in color) will be eliminated and some contouring of the graft will be done to fit the prepared envelope. The harvested SCTG will be placed at the extraction sites in a supra-periosteal partial dissection (pouch II technique) prepared at the buccal aspect without using vertical incisions and without flap elevation.
  Interventions: Other: SubEpithelial connective graft
- Atraumatic extraction (No Intervention): Extraction with Periotomes and Luxators keeping the buccal plate of bone intact

INTERVENTIONS:
Other: SubEpithelial connective graft — Connective tissue graft harvested from hard palate, to be placed buccal to extraction sockets in the intervention group
  Arms: SubEpithelial connective graft

SUMMARY:
This study will monitor the effect of soft tissue augmentation using sub-epithelial connective tissue graft buccal to extraction sockets in anterior maxilla in thin dento-alveolar phenotype; and will evaluate whether it will enhance the alveolar ridge contour and improve the gingival phenotype following atraumatic extraction compared with no treatment at all in terms of Ridge contour Preservation for future esthetically acceptable fixed prothesis.

DETAILED DESCRIPTION:
The aim of this study is to assess the alveolar ridge contour after soft tissue augmentation using sub-epithelial connective tissue graft buccal to fresh extraction sockets in patient with thin buccal bone, versus atraumatic extraction with no soft tissue augmentation.

Group A: Patients receiving atraumatic extraction with soft tissue augmentation by sub-epithelial connective tissue graft buccal to extraction sockets.

Group B: Patients receiving normal atraumatic extraction with no soft tissue augmentation

Clinical examination:

* Evaluation of the patient's general condition of the oral cavity, to make sure it complies with the criteria required to be enrolled in the study in terms of oral hygiene and pathological conditions.
* Evaluation of the buccal bone thickness using CBCT as diagnostic aid. (After CBCT if the patient was excluded because of thick buccal bone, he/she will be referred for implant placement)
* Evaluation of gingival phenotype before extraction using visual technique via periodontal probe.
* After patient enrollment, full mouth scaling to be done first and home oral hygiene measures to be done by patient. At the day of the surgery, immediately before extraction, an impression will be taken using alginate material and wax molded stock tray for recording the original ridge contour as the baseline data. casts will be made with dental extra hard stone.

Surgical procedure:

After administration of local anesthesia, the tooth will be extracted without raising flaps, as atraumatic as possible without disturbing the papillary tissues. After the extraction of the tooth, the socket will be carefully cleaned to excavate the granulation tissue in the marginal and apical regions.

Group A will receive atraumatic extraction and soft tissue augmentation using SCTG harvested from palatal tissue by single line incision technique blade will be oriented perpendicular to the palatal tissue surface. A single incision will be made down to the bone in a horizontal direction approximately 2 to 3 mm apical to the gingival margin of the maxillary teeth. A partial thickness dissection will then be made within the single incision, leaving an adequate thickness of the palatal flap intact to minimize the chance of sloughing of the overlying tissue. Careful manipulation of the graft with tissue forceps will be required and care must be taken to prevent compression or tearing of the graft.

The fatty tissue (yellow in color) will be eliminated and some contouring of the graft will be done to fit the prepared envelope. The harvested SCTG will be placed at the extraction sites in a supra-periosteal partial dissection (pouch II technique) prepared at the buccal aspect without using vertical incisions and without flap elevation. Sutures will be used to stabilize the graft in its desired place.

Pouch II technique:

A SCTG with a minimum thickness of 1.5 mm will be harvested from the palate. Following extraction, a full-thickness envelope flap will be created between the facial bone plate and the overlying gingiva. The SCTG will be inserted into the prepared envelope and secured with resorbable suture material. The apico-coronal dimension of the SCTG will be standardized throughout all the cases.

Group B will receive atraumatic extraction with no soft tissue augmentation.

(All patients assigned to the study will be referred to receive Prosthesis after treatment.)

ELIGIBILITY:
Inclusion Criteria:

* Adults from the age of 18 - 40 years
* Patients with non-restorable maxillary teeth/tooth indicated for extraction in the area from 2nd premolar to 2nd premolar
* Intact gingival tissue with at least 2mm keratinized tissue
* Buccal bone thickness should be 1mm or less assessed by CBCT before extraction
* Periodontally healthy patients
* Patients accepts to provide informed consent

Exclusion Criteria:

* Pregnant females.
* Smokers as smoking is a contraindication for any plastic periodontal surgery (Khuller, 2009).
* Handicapped and mentally retarded patients.
* Patients undergoing radiotherapy.
* Presence of systemic disease that would affect wound healing.
* Presence of active infection with soft tissue communication.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Buccal soft tissue contour | 6 Months
  Volumetric analysis using pre and post impressions and a digital software (V.Vanhoutte, et al. 2013) (Van Nimwegen, et al 2018). The soft tissue contours of the extraction sites will be assessed quantitatively. Impressions will be taken at 3 time-points, that is, before tooth extraction (baseline, T0) and 3 (T1), and 6 (T2) months after surgery. Plaster casts will be generated subsequently and digitised with a laser scanner. For the final analyses, CAD software is to be used to match the corresponding follow-up states (T1 to T2) with the baseline state (T0) and evaluate sections at defined positions with standardization of the apico-coronal dimension of SCTG.

SECONDARY OUTCOMES:
Gingival Thickness | 6 Months
  Gingival Thickness (GT) using Anesthetic Needle with a stopper (Paolantonio et al., 2002) will be measure at base line before extraction (T0), and during the follow up periods (T1 and T2)
Interdental Papilla height | 6 months
  height of papilla fill

CONTACTS AND LOCATIONS:
Overall Officials: Nourhan Gamal, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided